CLINICAL TRIAL: NCT06765837
Title: Effect of Low-Level Diode Laser Versus Active Oxygen Releasing Gel Application on Healing Outcome in Secondary Cleft Lip Correction
Brief Title: Comparison Between Low Level Laser Therapy and Active Oxygen Releasing Gel on Wound Healing Cleft Lip Patients
Acronym: LLLT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Hager Abd almonem, master's student at Faculty of dental medicine for girls and dentist at ministry of health, Faculty of Dental Medicine for Girls
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR SUR-106-1-C
Record Dates: First submitted 2024-12-29; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Cleft Lip
Keywords: Low level laser; cleft lip; scars; active oxygen releasing
MeSH Terms: conditions — Cleft Lip; Cicatrix

STUDY DESIGN:
Intervention Model Description: 3 groups underwent secondary repair cleft lip surgeries the first group subjected to low level laser after surgery the second group applied active oxygen releasing topical gel the third was a control group
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Low level laser therapy (Experimental)
  Interventions: Device: biolase laser
- active oxygen releasing gel (Experimental)
  Interventions: Drug: blue m gel
- control group (No Intervention)

INTERVENTIONS:
Device: biolase laser — after secondary cleft lip surgery to improve wound healing and prevent scar formation laser was used with group I and Gel was applied to Group II
  Arms: Low level laser therapy
Drug: blue m gel — active oxygen releasing gel was used after the secondary cleft lip repair surgery
  Arms: active oxygen releasing gel

SUMMARY:
the study was performed on secondary cleft lip scars

DETAILED DESCRIPTION:
the study aimed at comparing and Evaluation the effect of low-level diode laser and the effect of Active Oxygen releasing gel O3 (Blue-m gel) topical application on healing outcome in secondary cleft lip correction.

ELIGIBILITY:
Inclusion Criteria:

1. Age: can be done in any time after six months from the previous surgery if it severely disfiguring or in the preschool stage for children the time of surgery should be based on the severity of deformities
2. primary cleft lip repair was done
3. secondary lip repair with or without nose correction is indicated
4. the patient didn't undergo any surgeries procedures in the last 6 months

Exclusion Criteria:

1. previously subjected to secondary lip repair surgery.
2. syndromic cleft lip patient.
3. patient reporting abnormal reaction or scar healing in the previous surgery
4. smoking patients

Ages: 4 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Healing outcome of the wound is being measured by time | 6 months follow up
  measurements done by ultrasonography repeatedly , before and 1 week after surgery , 3 months after and 6 months after

CONTACTS AND LOCATIONS:
Overall Officials: Mohsena Ahmed, Study Director — lecturer of orthodontoics
Locations (1):
- Hager Abdelmonem Abdelaziz, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided